CLINICAL TRIAL: NCT04988659
Title: Total Exon Association Analysis of Femoroacetabular Impingement (FAI)
Brief Title: Analysis of Gene Expression in Femoroacetabular Impingement (FAI)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020533
Record Dates: First submitted 2021-06-25; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-06

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood from 100 patients with femoral acetabular impingement (FAI) was collected and DNA was extracted.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposures — Exposures

SUMMARY:
Femoral acetabular impingement (FAI) is a common disease of the hip joint. In this study, whole-genome sequencing was used to further explore the pathogenesis of this disease.

DETAILED DESCRIPTION:
Femoral acetabular impingement (FAI) is a group of chronic hip pain caused by the impact between the proximal femur and the edge of the acetabulum due to the anatomical abnormality of the hip joint, which damages the labrum and adjacent cartilage, and causes limited hip movement, especially limited flexion and internal rotation. However, the specific etiology of FAI is still unknown at present. The application of genome-wide, exon and transcription research methods to the study of hip impaction syndrome can uncover key differentially expressed genes and provide a theoretical basis for the study of FAI.

ELIGIBILITY:
Inclusion Criteria:

* The patient underwent preoperative imaging and was diagnosed with FAI. The patient complained of pain in the hip, hip, or thigh, and had a positive hip flexion impact test.

Exclusion Criteria:

* Patients with hip surgery history, hip osteoarthritis, necrosis of the femoral head, hip infection, hip dysplasia and other hip diseases.

Ages: 15 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Both patients were from Peking University Third Hospital and were diagnosed as Femoroacetabular impingement syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The patients were clinically diagnosed with FAI (femoral acetabular impingement) and underwent arthroscopic surgery, then clinical samples were collected. | The patient was diagnosed with FAI, and conservative treatment was ineffective for an average of 6 months.
  Peripheral blood from 100 patients with femoral acetabular impingement syndrome was collected and DNA was extracted.

CONTACTS AND LOCATIONS:
Overall Officials: yan xu, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No